CLINICAL TRIAL: NCT07010432
Title: The Role of the Amylin Analogue Cagrilintide in Bone Metabolism During Weight Loss in Postmenopausal Women With Obesity
Brief Title: The Role of the Amylin Analogue Cagrilintide in Bone Metabolism
Acronym: RAMBO
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9388-8175; U1111-1313-0864 (Other: World Health Organization (WHO)); 2024-517883-49 (Other: European Medical Agency (EMA))
Record Dates: First submitted 2025-05-30; First posted 2025-06-08 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — cagrilintide; semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cagrilintide (Experimental): Participants will receive once-weekly subcutaneous (s.c) injections of cagrilintide or placebo at stepwise doses every 4 weeks in a 16-week dose escalation period until target dose is achieved and maintained for 52 weeks as adjunct to a reduced calorie diet.
  Interventions: Drug: Cagrilintide; Drug: Placebo cagrilintide
- Semaglutide (Experimental): Participants will receive once-weekly s.c injections of semaglutide or placebo at stepwise doses every 4 weeks in a 16 week dose escalation period until target dose is achieved and maintained for 52 weeks as adjunct to a reduced calorie diet.
  Interventions: Drug: Semaglutide; Drug: Placebo semaglutide
- CagriSema (Experimental): Participants will receive once-weekly s.c injections of CagriSema (cagrilintide and semaglutide) or placebo at stepwise doses every 4 weeks in a 16 week dose escalation period until target dose is achieved and maintained for 52 weeks as adjunct to a reduced calorie diet.
  Interventions: Drug: Cagrilintide; Drug: Semaglutide; Drug: Placebo cagrilintide; Drug: Placebo semaglutide
- Placebo (Placebo Comparator): Participants will receive once-weekly s.c injection of placebo matched to semaglutide and cagrilintide for 68 weeks.
  Interventions: Drug: Placebo cagrilintide; Drug: Placebo semaglutide

INTERVENTIONS:
Drug: Cagrilintide — Participants will receive once-weekly cagrilintide subcutaneously.
  Arms: CagriSema; Cagrilintide
Drug: Semaglutide — Participants will receive once-weekly semaglutide subcutaneously.
  Arms: CagriSema; Semaglutide
Drug: Placebo cagrilintide — Participants will receive once-weekly placebo matched to cagrilintide subcutaneously.
  Arms: CagriSema; Cagrilintide; Placebo
Drug: Placebo semaglutide — Participants will receive once-weekly placebo matched to semaglutide subcutaneously.
  Arms: CagriSema; Placebo; Semaglutide

SUMMARY:
In this study we will investigate how the medicine cagrilintide affects bone health in women after menopause with obesity during weight loss, compared to treatment with placebo (the dummy medicine with no active substances) and semaglutide. The purpose is to examine whether cagrilintide can reduce the decline in bone mass associated to weight loss. Participants will either get cagrilintide, semaglutide, CagriSema (cagrilintide combined with semaglutide), or placebo. Which treatment participants get is decided by chance. Semaglutide is already approved for the treatment of overweight and obesity and can be prescribed by doctors. Cagrilintide and CagriSema are new medications currently under development for weight management. The study will last for about 79 weeks.

ELIGIBILITY:
Inclusion criteria

* Female.
* Post-menopausal at screening (defined as minimum 12 months of amenorrhea, high levels of follicular stimulating hormone (FSH) 16 - 130 international units per liter (IU/L), and low levels of anti-müllerian hormone (AMH) and inhibin B).
* Age 50-70 years (both inclusive) at the time of signing the informed consent.
* Body Mass Index (BMI) greater than or equal to >= 30.0 kilograms per square meter (kg/m^2).

Exclusion criteria

* Previous or current bone disease (e.g., osteoporosis, Paget's disease of bone, or bone cancer).
* Presence of disease affecting bone metabolism (e.g., diabetes mellitus, hyperparathyroidism, hyper or hypothyroidism, chronic kidney disease, celiac disease, or inflammatory diseases (e.g., psoriatic arthritis or ankylosing spondylitis)).
* Treatment with any medication affecting bone metabolism within 6 months prior to screening as judged by the investigator (e.g., anti-resorptive medication, anabolic medication, systemic hormone replacement therapy (HRT), or systemic corticosteroids).

Ages: 50 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-05-03 (Estimated); Study Completion 2028-05-03 (Estimated)

PRIMARY OUTCOMES:
Relative change in volumetric bone mineral density (vBMD) of the total hip assessed by quantitative computed tomography (QCT) | From baseline to end of treatment (week 68)
  Measured in percentage (%).

SECONDARY OUTCOMES:
Relative changes in vBMD of the lumbar 1 (L1) - L4 vertebrae assessed by QCT | From baseline to end of treatment (week 68)
  Measured in %.
Relative changes in vBMD of the radius assessed by QCT | From baseline to end of treatment (week 68)
  Measured in %.
Relative changes in vBMD of the L1 - L4 vertebrae assessed by QCT | From baseline to week 20
  Measured in %.
Relative changes in vBMD of the radius assessed by QCT | From baseline to week 20
  Measured in %.
Relative change in the Ki (bone turnover) of the femoral neck assessed by fluoride - positron emission tomography (PET) | From baseline to end of treatment (week 68)
  Measured in %.
Relative change in the Ki (bone turnover) of the femoral neck assessed by fluoride - PET | From baseline to week 20
  Measured in %.
Relative changes in C-terminal telopeptide of type I collagen (CTX-1) and procollagen type 1 N-terminal propeptide (P1NP) | From baseline to end of treatment (week 68)
  Measured in %.
Relative changes in CTX-1 and P1NP | From baseline to week 20
  Measured in %.
Relative changes in cortical thickness and porosity assessed by photon-counting computed tomography (PCCT) | From baseline to end of treatment (week 68)
  Measured in %.
Relative changes in trabecular thickness assessed by PCCT | From baseline to end of treatment (week 68)
  Measured in %.
Relative changes in number and separation of the femoral neck assessed by PCCT | From baseline to end of treatment (week 68)
  Measured in %.
Relative changes in L1-L2 vertebrae assessed by PCCT | From baseline to end of treatment (week 68)
  Measured in %.
Relative changes in radius assessed by PCCT | From baseline to end of treatment (week 68)
  Measured in %.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Steno Diabetes Center Copenhagen, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: http://novonordisk-trials.com